CLINICAL TRIAL: NCT03248570
Title: Phase 2 Open Label Study of Pembrolizumab in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC) With or Without DNA Damage Repair Defects
Brief Title: Pembrolizumab in Metastatic Castration Resistant Prostate Cancer (mCRPC) With or Without DNA Damage Repair Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16557; NCI-2017-02408 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA223484 (NIH)
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Castration Resistant Prostatic Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — pembrolizumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: After determination of DNA damage repair status, subjects will be assigned to one of two treatment groups:
  * Group 1 (DNA damage repair proficient group): Twenty-five subjects
  * Group 2 (DNA damage repair deficient group): Twenty-five subjects
  All subjects will receive pembrolizumab 200mg IV every 3 weeks until disease progression or unacceptable toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DNA damage repair proficient group (Experimental): Participants with mismatch repair (MMR) intact receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. If disease worsens while receiving pembrolizumab, participants may receive standard of care chemotherapy for 2-8 cycles
  Interventions: Drug: Pembrolizumab; Drug: Chemotherapy
- DNA damage repair defective group (Experimental): Participants with defective DNA repair receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. If disease worsens while receiving pembrolizumab, participants may receive standard of care chemotherapy for 2-8 cycles
  Interventions: Drug: Pembrolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab — All subjects will receive pembrolizumab 200mg IV every 3 weeks until disease progression or unacceptable toxicity.
  Other Names: KEYTRUDA; MK-3475
Drug: Chemotherapy — At time of progression, all subjects will also have the option of receiving taxane-based chemotherapy followed by repeat pembrolizumab for those who have a clinical response to chemotherapy. Chemotherapy regimen will be at the discretion of the treating physician, and may consist of docetaxel or cabazitaxel with or without a platinum agent (e.g. carboplatin). A minimum of 4 cycles and a maximum of 8 cycles of chemotherapy will be given.

SUMMARY:
This is a multicenter phase 2 open label study of pembrolizumab in patients with metastatic castrate resistant prostate cancer (mCRPC) with or without DNA damage repair defects.

DETAILED DESCRIPTION:
This is a multicenter phase 2 open label study of pembrolizumab in patients with metastatic castrate resistant prostate cancer (mCRPC) with or without DNA damage repair defects.

All subjects will receive pembrolizumab 200mg intravenously (IV) every 3 weeks until disease progression or unacceptable toxicity. The primary endpoint of the study is objective response rate (ORR) according to immune-mediated response criteria (irRC).

ELIGIBILITY:
Inclusion Criteria:

1. Documented histology of adenocarcinoma of the prostate.
2. Metastatic castration resistant prostate cancer with castrate-level testosterone (<50 ng/dL).

   a. Subjects must maintain a castrate-level testosterone during the study.
3. Disease progression defined by one or more of the following three criteria:

   1. Prostate-specific antigen (PSA) > 2.0 ng/mL and rising PSA by at least 2 consecutive measurements a minimum of 1-week apart.
   2. Soft tissue progression as defined by RECIST v1.1 criteria.
   3. Bone disease progression as defined by Prostate Cancer Clinical Trials Working Group 3 (PCWG3).
4. Have received prior secondary hormonal therapy including abiraterone, enzalutamide and/or apalutamide.
5. Be taking prednisone at a dose of ≤ 10mg/day, 7 days prior to starting treatment (Cycle 1, Day 1).
6. Be willing and able to provide written informed consent/assent for the trial.
7. Be >= 18 years of age on day of signing informed consent.
8. Patients must agree to have a tumor tissue biopsy at baseline, and there must be a lesion that can be biopsied with acceptable clinical risk as judged by the investigator.

   1. Patients with inconclusive DNA damage repair status testing on this baseline biopsy must have one of the following (per the investigator's discretion): (i) Sufficient archival tissue, or (ii) An additional biopsy attempt.
   2. Patients with previously identified homozygous deletion or deleterious germline or somatic mutation(s) in DNA damage repair gene(s) (such as BReast CAncer gene 1 (BRCA1) , BReast CAncer gene 2 (BRCA2), and ATM) identified in a Clinical Laboratory Improvement Amendments of 1988 (CLIA)-certified laboratory are allowed in Group 2. (i) Somatic mutation(s) in DNA damage repair gene(s) needs to be identified on the biopsy of a castration-resistant tumor site (ii) Archival FFPE tissue will be requested for determination of MSI (if not already assessed by gene sequencing) signature status.(iia) A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 10 slides containing unstained, freshly cut, serial sections must be available along with an associated pathology report before study enrollment. (iii) If archival FFPE tissue is unable to be obtained or is insufficient, patients will be required to undergo tumor tissue biopsy if feasible for determination of MSI signature status.
   3. Patients with germline mutation(s) in mismatch repair (MMR) gene(s) (i.e. Lynch syndrome),or have previously identified Microsatellite instability (MSI)-high tumor by Polymerase chain reaction (PCR) or MMR deficient tumor by Immunohistochemistry (IHC) are also allowed in Group 2. (i) Archival FFPE tissue will be requested for determination of Fanconi anaemia (FA)/BRCA signature status. (ia) A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 10 slides containing unstained, freshly cut, serial sections must be available along with an associated pathology report before study enrollment. (ii) If archival FFPE tissue is unable to be obtained or is insufficient, patients will be required to undergo tumor tissue biopsy if feasible for determination of FA/BRCA signature status.
9. If group 1 is not filled, patients may proceed onto treatment without the completion of tests for DNA repair status. Once group 1 is filled, patients cannot be enrolled onto the study or start treatment until DNA damage repair status is successfully determined for study group placement.

   a. Patients will be replaced if they have tissues that are not evaluable for DNA repair mutations
10. Patients must be willing to provide archival tissue from prior biopsy or surgery for prostate cancer, if available.

    a. A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 10 slides containing unstained, freshly cut, serial sections must be available along with an associated pathology report before study enrollment.
11. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
12. Patients must discontinue antiandrogen therapy (i.e. bicalutamide, flutamide, nilutamide) at least 4-6 weeks prior to registration with no evidence of PSA decline after washout.

    1. Bicalutamide: Washout period at least 6 weeks
    2. Flutamide and nilutamide: Washout period at least 4 weeks
13. Patients must discontinue therapies for mCRPC, with the exception of Gonadotropin-releasing hormone (GnRH) agent, for 14 days, with the exception of anti-androgens with which there may be a withdrawal PSA response.

    1. Prior chemotherapy is allowed if no progression of disease on chemotherapy.
    2. Prior treatment with sipuleucel-T, radium-223, or poly ADP-ribose polymerase (PARP) inhibitor (e.g. olaparib) is allowed.
    3. Tissue biopsy may be performed during washout period.
14. Demonstrate adequate organ function as defined as follows, all screening labs should be performed within 28 days of treatment initiation.

    1. Hematological: (i) Absolute neutrophil count (ANC): >= 1,500 /microliters (mcL) (ii) Platelets: >= 100,000 / mcL (iii) Hemoglobin: >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
    2. Renal: (i) Serum creatinine OR Measured or calculated a creatinine clearance (GFR can also be used in place of creatinine or CrCl): <=1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. Creatinine clearance should be calculated per institutional standard
    3. Hepatic: (i) Serum total bilirubin: <= 1.5 X ULN (ii) Aspartate Aminotransferase (AST) (SGOT) and Alanine Aminotransferase (ALT) (SGPT): <= 2.5 X ULN OR <= 5 X ULN for subjects with liver metastases (iii) Albumin: >= 2.5 mg/dL
    4. Coagulation: (i) International Normalized Ratio (INR) or Prothrombin Time (PT): <= 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or Partial Thromboplastin Time (PTT) is within therapeutic range of intended use of anticoagulants (ii) Activated Partial Thromboplastin Time (aPTT): <= 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
15. Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Significant liver metastasis.
2. Prior taxane-based chemotherapy with progressive disease on chemotherapy.

   1. Prior docetaxel for metastatic hormone sensitive prostate cancer is allowed, if no progression of disease on docetaxel as defined by RECIST v1.1 and PCWG3.
   2. Prior taxane-based chemotherapy (i.e. docetaxel or cabazitaxel with or without platinum agent) for mCRPC is allowed if no progression of disease on chemotherapy as defined by RECIST v1.1 and PCWG3.
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy >10mg/day or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
5. Has a known history of active Bacillus Tuberculosis (TB).
6. Hypersensitivity to pembrolizumab or any of its excipients.
7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., <= Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., <= Grade 1 or at baseline) from adverse events due to a previously administered agent.

   1. Note: Subjects with <= Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   2. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy <= 10 mg of prednisone/day for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has known history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-PD-L1, or anti-PD-L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (HBV) (i.e Hepatitis B surface antigen (HBsAg) reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
20. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Oh, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 3 | 1 | 4
  60-69 years old | 5 | 3 | 8
  70-79 years old | 6 | 5 | 11
  80-89 years old | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 11 | 20
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-Free Survival Rate (rPFS) at 6 Months
Description: The rPFS rate is defined as the proportion of participants still alive at 6 months starting from the first day of study treatment with pembrolizumab. Participants will be censored on the date of documented tumor progression according to the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines or death due to any cause at 6 months. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. The 6-month rPFS rate and the 95% confidence interval will be reported by study group.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
proportion of participants | 0.513 [0.296 to 0.888] | 0.63 [0.402 to 1.00]

2. Primary Outcome: Median Overall Radiographic Progression-free Survival (rPFS)
Description: The median overall radiographic progression free survival (rPFS) is defined as the time from the first day of study treatment with pembrolizumab to the date of documented radiographic tumor progression according to the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines or death due to any cause, whichever occurs first. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. The median time in months and the 95% confidence interval will be reported by study group.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
months | 10.43 [4.28 to NA] — The upper range of the confidence interval was calculated to be infinity | 7.89 [4.61 to NA] — The upper range of the confidence interval was calculated to be infinity

3. Secondary Outcome: Immune-related Progression-free Survival Rate (irPFS) at 20 Weeks
Description: The immune-related Progression Free Survival rate (irPFS) is defined as the proportion of participants still alive at 20 weeks from the first day of study treatment with pembrolizumab. Participants will be censored on the date of documented tumor progression according to the immune-related response criteria (irRC) for immune-related progression or death due to any cause at 20 weeks. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. The 20-week irPFS rate and the 95% confidence interval will be reported by study group.
Time Frame: Up to 20 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
proportion of participants | 0.513 [0.296 to 0.888] | 0.648 [0.421 to 0.998]

4. Secondary Outcome: Immune-related Progression-free Survival Rate (irPFS) at 28 Weeks
Description: The immune-related Progression Free Survival rate (irPFS) is defined as the proportion of participants still alive at 28 weeks from the first day of study treatment with pembrolizumab. Participants will be censored on the date of documented tumor progression according to the immune-related response criteria (irRC) for immune-related progression or death due to any cause at 28 weeks. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. The 28-week irPFS rate and the 95% confidence interval will be reported by study group.
Time Frame: Up to 28 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
proportion of participants | 0.513 [0.296 to 0.888] | 0.648 [0.421 to 0.998]

5. Secondary Outcome: Overall Progression-Free Survival Rate (PFS) at 20 Weeks
Description: The overall progression free survival rate (PFS) is defined as the proportion of participants still alive from the first day of study treatment with pembrolizumab at 20 weeks. Participants will be censored on the date of documented tumor progression using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines or death due to any cause at 20 weeks. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. The 20-week overall PFS rate and the 95% confidence interval will be reported by study group.
Time Frame: Up to 20 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
proportion of participants | 0.462 [0.257 to 0.83] | 0.556 [0.328 to 0.941]

6. Secondary Outcome: Overall Progression-Free Survival Rate (PFS) at 28 Weeks
Description: The overall progression free survival rate (PFS) is defined as the proportion of participants still alive from the first day of study treatment with pembrolizumab at 28 weeks. Participants will be censored on the date of documented tumor progression using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines or death due to any cause at 28 weeks. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. The 28-week overall PFS rate and the 95% confidence interval will be reported by study group.
Time Frame: Up to 28 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
proportion of participants | 0.462 [0.257 to 0.83] | 0.556 [0.328 to 0.941]

7. Secondary Outcome: Percentage of Participants Achieving Any Prostate Specific Antigen (PSA) Response
Description: The percentage of participants with a demonstrated PSA response will be reported for each group along with the 95% confidence interval.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
percentage of participants | 57.1 [28.9 to 82.3] | 58.3 [27.7 to 84.8]

8. Secondary Outcome: Percentage of Participants Achieving Any PSA Decline ≥ 50%
Description: The percentage of participants with a demonstrated PSA decline >= 50% will be reported for each group along with the 95% confidence interval.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
percentage of participants | 21.4 [4.7 to 50.8] | 41.7 [15.2 to 72.3]

9. Secondary Outcome: Number of Participants Reporting Any Pembrolizumab Treatment-related Adverse Events
Description: All participants will be evaluated for toxicity from the time of the first treatment with pembrolizumab. The number of participants with adverse events defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and categorized as having a possible, probable, or definite attribution to the administration of pembrolizumab from the start of treatment until 30 days after the end of treatment will be reported for each group.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 14 | 12
Participants | 11 | 11

10. Secondary Outcome: Median Time to Progression After Taxane-based Chemotherapy
Description: For participants who undergo taxane-based chemotherapy after progression on pembrolizumab followed by repeat pembrolizumab after chemotherapy, time from the first chemotherapy treatment to disease progression will be estimated in both study groups. Disease progression will be defined by confirmed PSA progression on two consecutive measurements at least 2 weeks apart, or radiographic progression by irRC. The Kaplan-Meier method will be used to estimate the median time to progression with 95% confidence interval by study group.
Time Frame: Up to 24 months
Population: data on not collected
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | DNA Damage Repair Proficient Group | DNA Damage Repair Defective Group
All-Cause Mortality (participants affected / at risk) | 8/14 | 8/12
Serious Adverse Events (participants affected / at risk) | 1/14 | 7/12
Other Adverse Events (participants affected / at risk) | 14/14 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DNA Damage Repair Proficient Group (N=14) | DNA Damage Repair Defective Group (N=12)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (2) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathologic femur fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DNA Damage Repair Proficient Group (N=14) | DNA Damage Repair Defective Group (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 6 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (9) | 6 (10)
Pain (General disorders) | 4 (6) | 3 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 7 (11) | 5 (10)
Urinary tract infection (Infections and infestations) | 1 (4) | 2 (4)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alkaline phosphatase increase (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 5 (5) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (9) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 1 (2)
Pelvic Pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study enrollment closed earlier than expected due to low enrollment. Some participants are still in follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT03248570/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03248570/ICF_000.pdf